CLINICAL TRIAL: NCT03250221
Title: Comparison of Robot-assisted Laparoscopic Myomectomy and Traditional Laparoscopic Myomectomy With Barbed Sutures
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: 106024-E
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Myomectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Robotic or laparoscopic myomectomy: Women who received robotic or laparoscopic myomectomy
  Interventions: Device: barbed sutures; Device: Vicryl@ suture

INTERVENTIONS:
Device: barbed sutures — Use of the barbed sutures for robotic or laparoscopic myomectomy
  Other Names: V-Loc
Device: Vicryl@ suture — Use of Vicryl@ suture for robotic or laparoscopic myomectomy

SUMMARY:
To elucidate the impact of barbed sutures on robotic myomectomy and laparoscopic myomectomy

DETAILED DESCRIPTION:
The aim of our study will be to elucidate the impact of the use of barbed sutures on robotic myomectomy and laparoscopic myomectomy

ELIGIBILITY:
Inclusion Criteria:

* All women who underwent robotic myomectomy and conventional laparoscopic myomectomy in the Department of Obstetrics & Gynecology of Far Eastern Memorial Hospital.

Exclusion Criteria:

* Open myomectomy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who underwent robotic myomectomy and conventional laparoscopic myomectomy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Abdominal drainage amount | 1 day
  Postoperative day 1 abdominal drainage amount

SECONDARY OUTCOMES:
Blood loss | 1 day
  Blood loss during surgeries
Surgical time | 1 day
  Surgical time

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Mou Hsiao, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

REFERENCES:
- [Background] Hsiao SM, Lin HH, Peng FS, Jen PJ, Hsiao CF, Tu FC. Comparison of robot-assisted laparoscopic myomectomy and traditional laparoscopic myomectomy. J Obstet Gynaecol Res. 2013 May;39(5):1024-9. doi: 10.1111/j.1447-0756.2012.02073.x. Epub 2013 Feb 4. PMID 23379670